CLINICAL TRIAL: NCT00768105
Title: A Randomized, Single-Blind, Placebo-Controlled, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Multiple Ascending Oral Doses of AZD1656 in Subjects With T2DM Treated With Insulin
Brief Title: To Evaluate Safety and Tolerability After Multiple Oral Doses of AZD1656 in Type 2 Diabetes Patients on Top of Insulin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: D1020C00014
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD1656
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Dose titration of oral suspension to a tolerable dose in 2-3 dose steps. Investigational product given twice daily for eight days.
  Arms: 1
Drug: Placebo — Dosing to match AZD1656
  Arms: 2

SUMMARY:
The purpose of this study is to assess safety and tolerability of AZD1656 after multiple repeated oral doses in patients with type 2 diabetes on top of insulin.

ELIGIBILITY:
Inclusion Criteria:

* Female with non child-bearing potential
* Diagnosed Diabetes Mellitus patients treated with insulin alone or insulin in combination with other anti-diabetic drugs. Stable blood sugar control indicated by no changed treatment within 3 months prior to study start.
* HbA1c below or equal to 11 % at screening (HbA1c value according to international DCCT standard)

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within two weeks before the first administration of the IP
* History of ischemic heart disease, stroke, transitorisk ischemic attack or symptomatic peripheral vascular disease
* Clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety variables (AE, BP, pulse, weight, plasma glucose, laboratory variables and ECG) | Blood samples taken repeatedly during 24 hours on study day sessions

SECONDARY OUTCOMES:
Pharmacokinetic variables | Blood samples taken repeatedly during 24 hours on study day sessions
Pharmacodynamic variables | Blood samples taken repeatedly during 24 hours on study day sessions

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Study Director — AstraZeneca R&D MÃ¶lndal; Marcus Hompesch, MD, Principal Investigator — Profil Institut for Clinical Research Inc.
Locations (1):
- Research Site, Chula Vista, California, United States